CLINICAL TRIAL: NCT02495142
Title: Psychosocial Issues and Bariatric Surgery
Acronym: LABS3
Status: Completed | Type: Observational
Sponsor: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Collaborators: Columbia University (Other); University of Pittsburgh (Other); Duquesne University (Other)
Responsible Party: Sponsor
Other Study IDs: 5R01DK084979-06 (NIH); NCT00582595 (obsolete NCT alias)
Record Dates: First submitted 2015-07-06; First posted 2015-07-13 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Eating Disorders; Bariatric Surgery Candidate; Depressive Disorder
MeSH Terms: conditions — Obesity; Feeding and Eating Disorders; Depressive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Bariatric surgery is associated with long-term weight loss, as well as short-term improvements in obesity-related medical comorbidities. However, a significant proportion of patients fail to lose sufficient weight, or experience significant weight regain. Although no robust predictors of response have been identified, pilot data that will be presented and reviewed suggest that surgery has profound effects on eating behaviors and psychosocial functioning, and that these factors may affect postoperative weight control.

The present investigation capitalizes on the Longitudinal Assessment of Bariatric Surgery (LABS) consortium to conduct an in-depth examination of the psychosocial aspects of surgery among a geographically, ethnically, and racially diverse sample of men and women undergoing bariatric surgery. This project unites experts in the areas of psychopathology, eating behaviors and quality of life to conduct a naturalistic study using state-of-the-art assessment tools; to document the relationships among psychosocial factors; and to examine psychosocial predictors of surgical outcomes.

DETAILED DESCRIPTION:
Primary Objective. Despite the obvious impact of bariatric surgery procedures on intake, no study to date has included a careful assessment of psychological factors, feeding patterns, energy intake and eating problems in this group of patients longitudinally. The Investigators believe that a careful examination of the structure of eating behavior and eating problems (e.g. vomiting) would be very helpful in guiding bariatric surgeons and dieticians who work with this group of patients in terms of dietary advice and recommendations, and with the prediction of eating problems and poor nutrient intake in the subgroup that develops such problems. This study involves prospective assessment of psychosocial outcomes of surgery by adding a supplemental battery to the LABS-2 assessment schedule. Conducting assessments at three of the LABS clinical sites assures the geographic, ethnic, and racial diversity of the sample, and hence enhances the potential to identify a subgroup or subgroups of patients susceptible to poor outcomes after surgery and the generalizability of study results.

This study would also include an evaluation of psychopathological and behavioral variables that might impact on weight loss and weight regain, and psychosocial complications post-operatively, as well as quality of life.

The overall goal of this study is to obtain detailed information that will allow a careful assessment of psychopathology, quality of life and eating behavior pre-surgically and at regular intervals for up to 7 years after the surgical intervention.

The Investigators believe that the instruments and procedures selected will allow a detailed examination of psychopathology, eating pathology and quality of life in detail.

The Investigators believe that the measures and tasks added at year 7 will allow the examination of theories of affect regulation, cognitive control, and reward processing in understanding postsurgical outcomes regarding pathological eating behavior and alcohol/substance use and their shared similarities as well as underlying neurobiological systems.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients who are at least 18 years of age and undergo bariatric surgery by a LABS certified surgeon.
* Previous enrollment in LABS-1 and LABS-2.
* BMI at baseline of greater than or equal to 35.

Exclusion Criteria:

* Informed consent not obtained
* Type 1 Diabetes Mellitus
* Unlikely to comply with follow-up protocol (ie: geographically inaccessible for study visits)
* Unable to communicate with local study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be approached for inclusion into LABS1 and LABS2 at the Sanford Surgery Department, Fargo ND, at the University of Pittsburgh Medical Center and at Cornell/Columbia Medical Center in New York. LABS3 Psychosocial participants will be selected from those individuals participating in LABS1 and LABS2.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Psychopathology as measured by the SCID | annually up to 7 years post bariatric surgery
  Structured Clinical Interview for DSM-IV, Patients Edition (SCID) will be administered to assess comorbid Axis I psychopathology.

SECONDARY OUTCOMES:
Change in Quality of life as measured by the IWQOL | annually up to 7 years post bariatric surgery
  Impact of Weight on Quality of Life Questionnaire: This is a 31-item, self-report, obesity-specific quality of life measure that will be utilized to assess quality of life.
Change in Quality of life as measured by the SF-36 | annually up to 7 years post bariatric surgery
  ShortForm-36: The SF-36 is a 36-item questionnaire that assesses functioning and quality of life as it relates to health status.
Change in Depression as measured by the BDI | annually up to 7 years post bariatric surgery
  Beck Depression Inventory: The BDI is a 21-item instrument that is widely used to assess depressive symptoms.
Change in Eating behaviors as measured by the EDE | annually up to 7 years post bariatric surgery
  Eating Disorder Examination: The diagnostic version of the EDE will be used as the primary measure of eating behavior and pathology.
Change in Impulse Control as measured by the SCID-ICD module | annually up to 7 years post bariatric surgery
  The impulse control module of the SCID will be administered to assess impulsive/compulsive disorders for participants.

OTHER OUTCOMES:
Affect regulation as measured by the DERS | 7 year post bariatric surgery
  Difficulties in Emotion Regulation Scale: The DERS is a 36-item self-report questionnaire that assesses six domains of emotion dysregulation and has been found to have acceptable internal consistency as well as adequate test-retest reliability and construct validity.
Affect regulation as measured by the AIM | 7 years post bariatric surgery
  Affect Intensity Measure:The AIM is a 40-item self-report measure of positive and negative emotional intensity and reactivity.
Impulsivity | 7 years post bariatric surgery
  UPPS-P Impulsive Behavior Scale: This is a 59-item self-report measure assessing five dimensions of impulsivity. Only the negative urgency and positive urgency subscales will be administered.
Behavioral inhibition as measured by the SPSRQ | 7 years post bariatric surgery
  Sensitivity to Punishment and Sensitivity to Reward Questionnaire: This is a 44-item self-report measure that is based on Gray's behavioral inhibition and activation motivational systems conceptualization, and assesses sensitivity to punishment and reward.
Temperament as measured by the ATQ | 7 years post bariatric surgery
  Effortful Control Scale of the Adult Temperament Questionnaire: This 19-item self-report measure assesses several components of dispositional effortful control, including attentional control (i.e., ability to voluntarily focus or shift attention), inhibitory control (i.e., ability to inhibit behavior), and activation control (i.e., ability to activate behavior as needed).
Cognitive Control as measured by the Go/No-Go Task | 7 years post bariatric surgery
  Go/No-Go Task: This computerized task assesses the capacity for suppressing previously reinforced responses.
Cognitive Control as measured by the Delay Discounting Task | 7 years post bariatric surgery
  Delay Discounting Task: Delay discounting tasks require participants to choose between receiving a larger amount of money after a delay versus receiving a smaller amount immediately.

CONTACTS AND LOCATIONS:
Overall Officials: James E. Mitchell, MD, Principal Investigator — Neuropsychiatric Research Institute
Locations (1):
- Neuropsychiatric Research Institute, Fargo, North Dakota, United States

REFERENCES:
- [Derived] Raatz SK, Johnson LK, Caliquary A, King WC, Kalarchian MA, Devlin MJ, Marcus MD, Mitchell JE. Reported nutrient intake over 7 years after Roux-en-Y gastric bypass in the Longitudinal Assessment of Bariatric Surgery-3 (LABS-3) psychosocial study. Surg Obes Relat Dis. 2020 Aug;16(8):1022-1029. doi: 10.1016/j.soard.2020.04.007. Epub 2020 Apr 22. PMID 32418771